CLINICAL TRIAL: NCT04484168
Title: Axial Ablation Versus Terminal Interruption of the Reflux Source (AAVTIRS): A Randomised Controlled Trial
Brief Title: Axial Ablation Versus Terminal Interruption of the Reflux Source
Acronym: AAVTIRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Hospital Galway (Other)
Collaborators: Stewart R Walsh (Unknown); Wael Tawfick (Unknown); Thomas A Aherne (Unknown); Mark Twyford (Unknown); Marie O'Shaughnessy (Unknown)
Responsible Party: Principal Investigator, Colum Keohane, Specialist Registrar in Vascular Surgery, University College Hospital Galway
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA2416
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Venous Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Terminal Interruption of the Reflux Source (TIRS (Active Comparator): These patients will have foam sclerotherapy of the veins in the immediate vicinity of their venous ulcer and thereafter be managed in compression bandaging and followed up fro 6 months or until the ulcer has healed
  Interventions: Procedure: Terminal Interruption of the Reflux Source
- Axial Ablation (Active Comparator): These patients will undergo endovenous ablation of the great or small saphenous veins, or other large superficial veins exhibiting significant reflux
  Interventions: Procedure: Axial Ablation

INTERVENTIONS:
Procedure: Terminal Interruption of the Reflux Source — Foam Sclerotherapy of veins in the immediate vicinity of the venous ulcer
  Arms: Terminal Interruption of the Reflux Source (TIRS
Procedure: Axial Ablation — Endovenous ablation of venous reflux in the main superficial veins of the leg
  Arms: Axial Ablation

SUMMARY:
This randomised trial aims to compare the effect on ulcer healing of different means of managing venous reflux in the lower limb. It is a non-inferiority trial comparing endovenous ablation of the axial (Saphenous and other large veins) veins of the lowere limb, versus terminal interruption of the reflux source (TIRS). For the purposes of this trial TIRS will be achieved using foam sclerotherapy of the distal tributaries in the immediate vicinity of the ulcer being treated.

ELIGIBILITY:
Inclusion Criteria

Primary or recurrent venous leg ulcer

Long or short saphenous vein reflux confirmed on ultrasound assessment, defined as retrograde flow lasting for >0.5 seconds

Ankle-Brachial pressure Index (ABI) ≥ 0.8 (if ulceration prevents ABI Toe-Brachial Index(TBI) ≥ 0.5 acceptable), or a palpable pulse

Ulcer size between 1 and 200 cm2

Patient suitable for full compression bandaging

Exclusion criteria Pregnancy (or breastfeeding and needing to feed within 48 hours of treatment)

Active infection of ulcer, or infection within the last two weeks

Leg ulcer of non-venous aetiology as determined by clinical assessment

Isolated perforator vein reflux only

Evidence of deep venous insufficiency or thrombosis

Known hypersensitivity to Sotradecol or similar sclerosants

Previous inability to tolerate compression bandages

Presence of any contraindications for the use of compression bandages:

Absence of a palpable pulse, and Ankle Brachial Index (ABI) <0.8

Decompensated congestive cardiac failure (NYHA Class IV)

Known hypersensitivity to any of the component materials

Patients unable to provide informed consent

Patients attending the leg ulcer clinic already will be excluded from enrolment with the same ulcer but will be eligible to enrol with a contralateral ulcer. Recurrent ipsilateral ulcers will not be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Ulcer healing | 6 months
  The main outcome measure is the proportion of ulcers which have healed within the follow up period

SECONDARY OUTCOMES:
Ulcer Healing | 3 months
  The proportion of ulcers healed at three months
Reduction in ulcer size | 6 months
  The absolute reduction in ulcer size in square cm
Relative Reduction in ulcer size | 6 months
  Reduction in ulcer size as a percentage of original ulcer area
Wound Progress | 6 months
  Progress in Wound regeneration as indicated by changes in Bates-Jensen Wound Assessment Tool (BWAT)
Change in overall venous disease | 6 months
  Monthly change in Venous Clinical Severity Score
Change in Venous disease related quality of Live | 6 months
  Changes in Charing Cross Venous Ulcer Quesionnaire score from randomisation to exit from the study

CONTACTS AND LOCATIONS:
Overall Officials: Colum R Keohane, MB,BCh,BAO, Principal Investigator — UCH Galway and NUI Galway
Locations (1):
- Roscommon Unversity Hospiral, Roscommon, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cr K, D W, M T, T A, W T, Sr W. Axial Ablation versus Terminal Interruption of the Reflux Source (AAVTIRS): A Randomised Controlled Trial. Vasc Endovascular Surg. 2024 Nov;58(8):805-812. doi: 10.1177/15385744241265750. Epub 2024 Jul 21. PMID 39034428
- [Derived] Keohane CR, Westby D, Twyford M, Ahern T, Tawfick W, Walsh SR. Axial ablation versus terminal interruption of the reflux source (AAVTIRS): a randomised controlled trial. Trials. 2022 Jun 10;23(1):483. doi: 10.1186/s13063-022-06440-4. PMID 35689289